CLINICAL TRIAL: NCT01819662
Title: Stratified Management of Patients With Pacemakers
Brief Title: Optimised Pacing Program
Acronym: OPT-pace
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Leeds (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, KK Witte, Principle Investigator, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: NIHR-CS-012-032
Record Dates: First submitted 2013-03-24; First posted 2013-03-27 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Pacemaker Complication; Congestive Heart Failure
Keywords: Pacemaker, heart failure, hospitalisation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard management (Placebo Comparator): No echocardiogram
  Interventions: Other: Standard management
- Enhanced standard management (Active Comparator): Echocardiogram performed, with results to GP
  Interventions: Other: Enhanced standard management
- Optimised heart failure management (Active Comparator): Echocardiogram, followed by referral to comprehensive heart failure program for those with left ventricular dysfunction
  Interventions: Other: Optimised heart failure management

INTERVENTIONS:
Other: Enhanced standard management — Echocardiogram followed by letter to GP about results.
  Arms: Enhanced standard management
Other: Optimised heart failure management — Echocardiogram followed by referral to comprehensive heart failure service for those with left ventricular dysfunction
  Arms: Optimised heart failure management
Other: Standard management — Usual care
  Arms: Standard management

SUMMARY:
Permanent pacemakers are a common treatment for slow heart beats. In the UK 300,000 people have a pacemaker, and each year another 36,000 receive them. All of these patients are usually seen yearly to have their device checked. However, pacemaker technology is now very reliable, batteries last well over 5 years, and many patients require their pacemaker only occasionally as a back-up. Each visit costs around £200 such that pacemaker follow-up cost the NHS around £50million per year. Most visits involve checking the battery and the leads which, in the absence of symptoms might be unnecessary.

Pacemaker patients are at risk of developing other problems including heart failure which puts them at higher risk of hospitalisation and death. For those under follow-up, no mechanism exists to identify whether they might have heart failure, and for those receiving new implants, it is unclear which will go on to develop heart failure. Also, whether optimal heart failure treatment with a multidisciplinary team reduces the chances that they will be hospitalised is also unproven.

Our study therefore has three main aims: 1) based on pacing indications and patient factors, to identify which patients are likely to develop complications and therefore which patients could be seen less frequently; 2) to validate and refine a simple risk score to help identify which patients in pacing clinic should undergo screening for heart failure; and 3) to establish whether such screening and subsequent optimisation of those with heart failure is clinically and cost-effective for reducing hospitalisation and death.

DETAILED DESCRIPTION:
Permanent pacemaker implantation is a safe, life-prolonging and cost-effective treatment for bradycardia. An estimated 300,000 people in the UK have a pacemaker and there are 36,000 new implants per year. Complications from pacemaker implantation occur in 5-15% of patients, mostly in the first six weeks. After six months new problems are very rare. Clinic follow-up of patients with a PPM usually occurs at six weeks, three months and then annually to monitor battery performance. Reprogramming is rarely required, and batteries reliably last at least five years. The tariff for pacemaker follow-up is £200 costing the National Health Service (NHS) £50 million per year.

The commonest and most under-recognised long-term complication of pacemaker implantation is pacemaker-related chronic heart failure (CHF) due to left ventricular systolic dysfunction, seen in up to 50% of patients. Published data examining the incidence and associations of pacemaker-related cardiac dysfunction consist of retrospective cross-sectional analyses or data taken from other studies rather than a-priori planned analyses. Our unique pilot data in almost 500 patients show that cardiac dysfunction is present in 40% of all pacemaker patients and confirm previous suggestions that it is more common in patients with an underlying predisposition, for example cardiovascular co-morbidities (including diabetes mellitus), with high rates of pacing and atrial fibrillation. Our data also demonstrate that patients with cardiac dysfunction and a pacemaker are not usually taking optimal medical therapy for their heart failure and suffer a 13% annual combined heart failure hospitalisation or death rate (compared to 6% in pacemaker patients without cardiac dysfunction, and ~8% in patients with CHF attending the Leeds Integrated Heart Failure Service). However, since patients with pacemakers were often excluded from the large studies of medical (and device) therapy of CHF, it is unclear whether optimisation of medical (and pacemaker) therapy in patients with pacemaker-related cardiac dysfunction can reduce mortality and hospitalisation. Pilot data from our clinic in 25 patients with a pacemaker and CHF, show that optimised medical therapy can lead to similar improvements in cardiac function as in CHF patients without a pacemaker.

The present project therefore includes three distinct, but closely related, work packages which will answer three questions;

1. in patients receiving their first pacemaker, which clinical and pacing variables predict short, medium and long-term complications and is it therefore feasible, safe and cost-effective to individualise follow-up intervals;
2. can we confirm and validate our previous observation that a model consisting of simple clinical and pacing variables identifies pacemaker patients at higher risk for cardiac dysfunction during a pacemaker-follow-up appointment and;
3. does applying our risk model with subsequent optimisation of medication and pacemaker programming within a multidisciplinary heart failure service in those with heart failure lead to cost effective and clinically relevant reductions in mortality and hospitalisation?

ELIGIBILITY:
Inclusion Criteria:

* Pacemaker implantation

Exclusion Criteria:

* Dementia, unwilling to fill in quality of life questionnaires, unwilling to sign consent form

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1793 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Combined hospitalisation and mortality | 3 years

SECONDARY OUTCOMES:
Predictors of complications from pacemaker implantation | 3 years

OTHER OUTCOMES:
Predictors of cardiac dysfunction in pacemaker patients | 1-3 years
  Who will develop cardiac dysfunction after permanent pacemaker implantation? Who under follow-up has cardiac dysfunction and how can it be identified?

CONTACTS AND LOCATIONS:
Overall Officials: Klaus K Witte, MD, Principal Investigator — University of Leeds
Locations (3):
- United Kingdom (3):
  - Bradford Hospitals NHS Foundation Trust, Bradford, Yorkshire
  - Harrogate Hospital Foundation Trust, Harrogate, Yorkshire
  - Leeds General Infirmary, Leeds

REFERENCES:
- [Derived] Paton MF, Gierula J, Jamil HA, Straw S, Lowry JE, Byrom R, Slater TA, Fellows AM, Gillott RG, Chumun H, Smith P, Cubbon RM, Stocken DD, Kearney MT, Witte KK. Echocardiographic screening for heart failure and optimization of the care pathway for individuals with pacemakers: a randomized controlled trial. Nat Med. 2024 Nov;30(11):3303-3309. doi: 10.1038/s41591-024-03265-3. Epub 2024 Sep 19. PMID 39300290
- [Derived] Paton MF, Gierula J, Jamil HA, Lowry JE, Byrom R, Gillott RG, Chumun H, Cubbon RM, Cairns DA, Stocken DD, Kearney MT, Witte KK. Optimising pacemaker therapy and medical therapy in pacemaker patients for heart failure: protocol for the OPT-PACE randomised controlled trial. BMJ Open. 2019 Jul 17;9(7):e028613. doi: 10.1136/bmjopen-2018-028613. PMID 31320354